CLINICAL TRIAL: NCT01429493
Title: Biological Image Guided Antalgic Stereotactic Body Radiotherapy of Bone Metastases: a Randomized Phase II/III Trial
Brief Title: Biological Image Guided Antalgic Stereotactic Body Radiotherapy of Bone Metastases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/541
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Bone Metastases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional radiotherapy (Active Comparator)
  Interventions: Radiation: Conventional Radiotherapy
- Biological image-guided radiotherapy with conventional dose. (Experimental)
  Interventions: Radiation: Biological image-guided radiotherapy with conventional dose.
- Biological image-guided SBRT with dose-escalation. (Experimental)
  Interventions: Radiation: Biological image-guided SBRT with dose-escalation.

INTERVENTIONS:
Radiation: Conventional Radiotherapy — Conventional radiotherapy will be used (8 Gy/ 1 fraction).
  Arms: Conventional radiotherapy
Radiation: Biological image-guided radiotherapy with conventional dose. — Biological image-guided radiotherapy on the positron emitting tomography (PET) positive lesion with conventional dose (8Gy/ 1 fraction) will be used.
  Arms: Biological image-guided radiotherapy with conventional dose.
Radiation: Biological image-guided SBRT with dose-escalation. — Biological image-guided stereotactic body radiotherapy (SBRT) with dose-escalation on the PET positive lesion will be used.
  Arms: Biological image-guided SBRT with dose-escalation.

SUMMARY:
In various common cancers, the skeleton is a preferred site of metastasis. These bone metastases are the most common cause of cancer-related pain, which significantly impair quality of life. It is postulated that the clinical target volume (CTV) of painful bone metastases consists of cancer cells and tumor-associated host cells: the tumor-host ecosystem. Advances in biological imaging (positron emitting tomography PET) might allow us to selectively identify the tumor-host ecosystem within the anatomical boundaries of a bone metastasis. These findings suggest the potential of intentionally non-homogenous dose escalation (dose painting by numbers) to improve pain control. The hypothesis is that fluorodeoxyglucose positron emitting tomography (FDG-PET) can detect the intra-bone metastasis regions confined with tumor-associated host-cell compartments responsible for metastasis-related pain. The primary objective is to improve pain control with biological image-guided stereotactic body radiotherapy compared to conventional radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Painful bone metastasis of solid tumors
* Pain score minimum of 2 on a scale of 10
* A maximum number of painful bone metastases: 3 or more
* Life expectancy > 3 months
* Age minimum 18 years old
* Signed informed consent

Exclusion Criteria:

* Tumor histology (renal cell and melanoma vs. other solid tumors)
* VAS pain score (<5 vs. 6-10).
* Bisphosphonate use (yes vs. no)
* Opioid analgesics (yes vs. no)
* Corticosteroid use (yes vs. no)
* Spine vs non-spine localisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Level of pain response 1 month after radiotherapy | 1 month after radiotherapy
  Pain is measured with the visual analogue scale. Response is scored in accordance to the guidelines of the international consensus on palliative radiotherapy.

SECONDARY OUTCOMES:
Quality of life 1 month after radiotherapy. | 1 Month after radiotherapy
  Quality of life 1 month after radiotherapy measured with the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Bone Metastases Module (QLQ-BM22).

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - Ghent University Hospital, Ghent

REFERENCES:
- See also: Related Info — http://www.uzgent.be